CLINICAL TRIAL: NCT02643901
Title: The Single-Dose Tolerability and PK/PD Study of Recombinant (Expressed by Pichia Pastoris) Human Serum Albumin/Human Granulocyte-Colony Stimulating Factor(I) Fusion Protein for Injection (GW003) in Healthy Subjects
Brief Title: Tolerability and Pharmacokinetics(PK)/Pharmacodynamics(PD) Study of GW003 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu T-Mab Biopharma Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tmab-GW003-NP-03
Record Dates: First submitted 2015-11-30; First posted 2015-12-31 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2016-09

CONDITIONS: Chemotherapy-induced Neutropenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Ic-GW003 150ug/kg 4-8subjects (Experimental): Biological/Vaccine:GW003 freeze-dried powder single SC injection
  Interventions: Biological: GW003
- Ic-GW003 300ug/kg 6-8subjects (Experimental): Biological/Vaccine:GW003 freeze-dried powder single SC injection
  Interventions: Biological: GW003
- Ic-GW003 500ug/kg 6-8subjects (Experimental): Biological/Vaccine:GW003 freeze-dried powder single SC injection
  Interventions: Biological: GW003
- Ic-GW003 650ug/kg 6-8subjects (Experimental): Biological/Vaccine:GW003 freeze-dried powder single SC injection
  Interventions: Biological: GW003
- Ic-GW003 850ug/kg 6-8subjects (Experimental): Biological/Vaccine:GW003 freeze-dried powder single SC injection
  Interventions: Biological: GW003

INTERVENTIONS:
Biological: GW003 — single SC injection

SUMMARY:
This study is designed to access the tolerability and Pharmacokinetic/Pharmacodynamic (PK/PD) of single subcutaneous (SC) injection of GW003 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* 18 years to 45 years,Healthy male and female subjects.in the same dose group,the age difference between in 10 years
* At least 50kg weight,BMI between 19 and 25kg/m2
* No tobacco, alcohol and other bad habits
* No history of drug allergy and biological agents allergy and other allergies
* Not used biological agents and other drugs within three months before participated in this test
* Not participated in other test or donated blood within three months before participated in this test
* The medical history、physical examination、laboratory examination is normal or slightly abnormal
* Subjects can obey the clinical trial protocol
* Subjects, who are willing to follow the study protocol and provide written informed consent voluntarily.

Exclusion Criteria:

* History of severe system disease(especially with the spleen swelling, adult respiratory distress syndrome and exudative pneumonia or sickle red blood cell anemia history)
* History of drug allergy and biological agents allergy and other allergies
* Subjects have used any long discharge period drugs will affect the present study within 3 months or are using drugs now
* Subjects not to take effective contraceptive measures or have a family planning within one year， Pregnancy or nursing women
* Subjects accepted major surgery 4 weeks before drug administration
* Subjects vaccinated live vaccine 3 months before drug administration
* Subjects with the history of drug abuse 5 years before drug administration
* As the subjects participated 3 times or more than 3 times drug clinical trials within 1 year or as the subjects participated any drug clinical trial or donated blood within 3 months
* Clinical and laboratory examination results is abnormal and have clinical significance
* Subjects with poor compliance or have any unfavorable factors to participate in this test
* Subjects can not complete the research
* The researchers and their family members.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2015-09; Primary Completion 2016-10-10 (Actual); Study Completion 2016-10-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | up to day 21
  To evaluate the safety and tolerance of single SC injection of GW003 in healthy subjects.

SECONDARY OUTCOMES:
Frequency of subjects with Anti-GW003 antibody | up to 6 months after the trial
  anti-GW003 was detected pre-dose and at the last visit,if there exist positive anti-GW003 antibody, another detected should be conducted 6 months after the trial.
half-life(consist of distribution and elimination half-life) for GW003 | up to day 14
area under the concentration-time curve(AUC) for GW003 | up to day 14

CONTACTS AND LOCATIONS:
Overall Officials: Qi Junyuan, doctor, Principal Investigator — Tianjin Hematonosis Hospital
Locations (1):
- Tianjin Hematonosis Hospital, Tianjin, Tianjin Municipality, China